CLINICAL TRIAL: NCT03655483
Title: A Single Arm，Multicenter， Phase II Clinical Study to Evaluate the Efficacy and Safety of GLS-010 Injection in the Treatment of Recurrent or Refractory Classical Hodgkin's Lymphoma
Brief Title: Study of GLS-010 Injection in the Treatment of Classical Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangzhou Gloria Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH-S001-04
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Classical Hodgkin's Lymphoma
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLS-010 (Experimental): GLS-010
  Interventions: Drug: GLS-010

INTERVENTIONS:
Drug: GLS-010 — Full-human anti-pd-1 monoclonal antibodies
  Other Names: Full-human anti-pd-1 monoclonal antibodies

SUMMARY:
Patients with refractory cHL. Patients will be treated with GLS-010

DETAILED DESCRIPTION:
Open, uncontrolled, multi-center, phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who met all the criteria below could be selected for the study:

  1. Willingness to participate in the clinical trial. Provide written informed consent prior to any study-specific screening procedures. Willingness and capability to comply with the requirements of the study;
  2. Male or female, Age between 18 and 70 years old (margin included) on the day of signing informed consent.
  3. Histologically confirmed diagnosis of cHL(classical Hodgkin Lymphoma);
  4. Relapsed or refractory classical Hodgkin Lymphoma patients after 2 or more lines of therapies( Relapsed cHL patients are defined as patients with new lesion found at primary site or other sites after achieving a complete response after the last treatment; refractory cHL is defined as patients achieve a less than complete response or partial response after the last treatment）and at least one of the following condition is in accordance with:

     1. Participant has failed to achieve a response after treatment with autologous stem cell transplant (auto-SCT) or relapsed after achieving a response.
     2. Participant has failed to achieve a response to, progressed after, or be ineligible for autologous stem cell transplant (auto-SCT)
  5. Based on Lugano 2014, at least one bi-dimensional measurable Lymph node lesion with minimum measurement of > 15 mm or an extranodal lesion with minimum measurement of > 10 mm in the longest diameter of cross-sectional areas in CT test, plus positive on Fluorodeoxyglucose-positron tomography（FDG-PET）.
  6. Paraffin embedding sample or biopsy sample available during screening;
  7. Must have ECOG performance status of 0 or 1
  8. Has a predicted survival period ≥ 12 weeks;
  9. Demonstrate adequate organ and hematopoietic function as defined below:

     1. Hemoglobin ≥8.0 g/dL
     2. Absolute neutrophil count (ANC) ≥1000 /mcL
     3. Platelets ≥75,000 / mcL
     4. Serum total bilirubin ≤ 1.5 X ULN
     5. AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
     6. Serum creatinine OR ≤1.5 X upper limit of normal (ULN)
     7. International Normalized Ratio (INR) or Prothrombin Time (PT)≤1.5 X ULN unless subject is receiving anticoagulant therapy, then as long as coagulation parameter (PT /INR or Activated Partial Thromboplastin Time (aPTT) , or anti-Xa factor )is within therapeutic range of intended use of anticoagulants.
  10. Since signing the ICF, female or male subjects of childbearing potential should be willing to use an adequate method of contraception with the spouse for the course of the study through 5 months after the last dose of study medication.

Exclusion Criteria:

* Subjects who met the following criteria were not eligible for the study:

  1. Nodular lymphocytes is confirmed as primary Hodgkin lymphoma or grey zone lymphoma.
  2. Has known active central nervous system (CNS) metastases.
  3. Has undergone allogeneic hematopoietic stem cell transplantation.
  4. Has undergone autologous stem cell transplantation within 100 days prior to the first dose of study drug.
  5. Grade 3 or 4 congestive heart failure (New York Heart Association (NYHA)), unstable angina pectoris, poorly controlled arrhythmias(including male QTc intervals≥ 450 ms, female QTc intervals≥ 470 ms, QTc intervals calculated by Formula Fridericia), acute ischemia on ECG or myocardial infarction within 6 months prior to screening.
  6. Patients with any autoimmune disease, i.e., but not limited to, interstitial pneumonia, uveitis, enteritis,hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism (hypothyroidism without clinical symptoms or caused by radiotherapy and chemotherapy can be included); Patients with vitiligo or asthma CR in Childhood, not requiring any intervention in adulthood are permitted to enroll.; patients with asthma requiring a bronchiectasis intervention are not permitted to enroll.
  7. Subjects that requires systemic corticosteroids (Dose equivalent to or above 10 mg prednisone daily) or other immunosuppressive medications;
  8. Has received a live anti-tumor vaccine, or anti-tumor treatment with immunostimulation within 4 weeks prior to pre-screening.
  9. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti CTLA-4 antibody (including Ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
  10. Presence of other active cancers within 5 years prior to enrollment. Patients with cervical carcinoma in situ/ cured skin basal cell carcinoma who have received definitive adequate treatment are eligible.
  11. Participants with active viral hepatitis (positive HepB sAg and/or positive HepB core Ab with positive HepB DNA> 103copies/mL, or positive HepC antibody), or syphilis positive.
  12. Has a known Human Immunodeficiency Virus (HIV) infection, or other acquired and congenital immune deficiency diseases, or history of organ transplant.
  13. Has history of active TB infection within 1 year prior to enrollment. (Suspected TB infection patient needs chest X-ray, sputum examination and clinical symptom for conformation. Patients with active TB infection should be excluded even if cured.)
  14. Subject that requires systematic treatment for active infection, unexplained fever> 38.5°C prior to the first dose of study drug during screening( Subjects that has tumor related fever could be included while confirmed by the investigator.)
  15. History of allergic reactions attributed to any macromolecular protein preparation/monoclonal antibody, or any other composition of the study drug.
  16. Investigational drug therapy outside of this trial during or within 4 weeks prior to GLS-010.
  17. Has had prior chemotherapy, radiation therapy, targeted small molecule therapy or major surgery within 4 weeks prior to the first dose of study drug; who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent (alopecia excluded)
  18. Has history of Interstitial Lung Disease or non-infectious pneumonitis (Patients caused by radiotherapy are eligible.)
  19. Has history of alcoholism or drug abuse within 1 year;
  20. Has clear history of neurological or mental disorders, i.e. epilepsy, dementia, and poor compliance.
  21. Has received an anti-infection vaccine within 4 weeks prior to the first dose of study drug (i.e. Influenza virus vaccines, HPV vaccines). Any live vaccines are not allowed during the study.
  22. Pregnancy or lactation.
  23. Other conditions that do not permit compliance with the protocol, evaluated by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2018-08-24 (Actual); Primary Completion 2021-04-11 (Estimated); Study Completion 2022-04-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 2 months
  Based on an independent image assessment board

SECONDARY OUTCOMES:
PFS | 8 weeks
  meaningful benefit in PFS based on Lugano 2014
OS | within 3 years of last patient enrolled
  Overall survival
DCR | 8 weeks
  meaningful benefit in DCR based on Lugano 2014
DOR | 8 weeks
  meaningful benefit in DOR based on Lugano 2014
TTR | 8 weeks
  meaningful benefit in TTR based on Lugano 2014

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute; Yuqin Song, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (5):
- China (5):
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - Hunan Cancer Hospital, Changsha, Hunan
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Peking University Cancer Hospital & Institute, Beijing

REFERENCES:
- [Derived] Kan S, Bai H, Liu H, Cui J, Ke X, Zhang H, Liu L, Yan D, Jiang Y, Zang A, Qi J, Wang L, Liu Z, Xu B, Zhang Y, Zhang Z, Zhao X, Hu C, Yang S, Zhou H, Shi J, Shao Z, Xiang Y, Lin N, Zhang M. Long-term follow-up of zimberelimab in relapsed or refractory classic Hodgkin lymphoma: Insights from the phase Ⅱ YH-S001-04 clinical trial. Leuk Res. 2025 Feb;149:107633. doi: 10.1016/j.leukres.2024.107633. Epub 2024 Nov 26. PMID 39799811
- [Derived] Lin N, Zhang M, Bai H, Liu H, Cui J, Ke X, Zhang H, Liu L, Yan D, Jiang Y, Zang A, Qi J, Wang L, Liu Z, Xu B, Zhang Y, Zhang Z, Zhao X, Hu C, Yang S, Zhou H, Shi J, Shao Z, Xiang Y, Zhu J, Song Y, Zhu J. Efficacy and safety of GLS-010 (zimberelimab) in patients with relapsed or refractory classical Hodgkin lymphoma: A multicenter, single-arm, phase II study. Eur J Cancer. 2022 Mar;164:117-126. doi: 10.1016/j.ejca.2021.07.021. Epub 2021 Aug 27. PMID 34462189